CLINICAL TRIAL: NCT04303442
Title: A Prospective Endoscopic Study of the Presence, Type and Size of Corona Mortis in 300 Patients Undergoing Total Extraperitoneal (TEP) Inguinal Hernia Repair Procedures
Brief Title: Corona Mortis in Patients Undergoing TEP for Inguinal Hernia
Status: Completed | Type: Observational
Sponsor: Sofia Med Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 207
Record Dates: First submitted 2020-03-08; First posted 2020-03-11 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Inguinal Hernia; Pelvic Fracture; Acetabular Fracture; Bleeding
Keywords: Corona Mortis; TEP; Inguinal Hernia; Laparoscopic Surgery; Anatomy; Inguinal region anatomy; Bleeding
MeSH Terms: conditions — Hernia, Inguinal; Hip Fractures; Hemorrhage | interventions — tetraethylpyrazine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing TEP: Patients diagnosed with unilateral or bilateral primary and/or recurrence inguinal hernia undergoing Total Extraperitoneal laparoscopic hernia repair.
  Interventions: Procedure: TEP

INTERVENTIONS:
Procedure: TEP — Total extraperitoneal laparoendoscopic hernia repair with one or three skin incisions.

SUMMARY:
This study aim to describe the presence, type and size of Corona mortis (CMOR) in patients undergoing total extraperitoneal (TEP) inguinal hernia repair procedures. This study also aim to describe the preperitoneal vascular anatomy of inguinal area and provide in vivo knowledge about CMOR.

DETAILED DESCRIPTION:
Corona mortis is classically defined as the arterial and/or venous vascular anastomosis between the obturator artery and external iliac artery (most commonly the inferior epigastric artery) that crosses the posterior aspect of the superior ramus of the symphysis pubis. It runs along the posterior aspect of the superior pubic ramus and its laceration can prove life threatening in trauma cases or in scheduled operations.

CMOR is clinically important due to the potential risk of bleeding in pelvic fractures, pelvic and acetabular operations, surgery for urinary incontinence, oncologycal pelvic dissections and laparoscopic hernia repair. It requires special interests from different surgical branches, such as orthopedics, oncologic surgery, urogynecology and general surgery. Vascular anatomy of retropubic area, especially CMOR, should be kept in mind by surgeons performing laparoscopic surgery for hernia repair. In literature, the anatomical data have usually been come from studies performed on cadavers. The aim of this study was to provide in vivo knowledge about the presence, type (venous and/or arterial) and size of CMOR in patients who underwent TEP repair.

300 patients will undergo TEP procedure for unilateral or bilateral inguinal hernias. TEP procedures will be performed with three ports and one or three skin incisions. The presence and type of CMOR will be evaluated, and picture will be made. The size of the CMOR will be defined with ruler inserted true the 10 mm port.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed primary or recurrence unilateral or bilateral inguinal hernia
* Age between 18 and 90;

Exclusion Criteria:

* Patients who prefer other surgical approach than TEP

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients male and female, undergoing TEP inguinal hernia repair.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Presence of CMOR | Intraoperative
  Evaluation of presence of Corona mortis in each hemipelvis examined. For unilateral hernias - one hemipelvis, in bilateral - two hemipelvices.
Type CMOR | Intraoperative
  Evaluation of the type of Corona Mortis - Arterial, Venous or both types, in each hemipelvis
Size of CMOR | Intraoperative
  Evaluation of size of Corona Mortis in mm., measured with ruler.

CONTACTS AND LOCATIONS:
Locations (1):
- Sofiamed Hospital, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No